CLINICAL TRIAL: NCT05098353
Title: Program to Study the Experience of Using Seroquel ® in Patients With Bipolar Disorder of the First and Second Types in Remission With Signs of Impaired Impulse Control
Brief Title: Seroquel ® in Patients With Bipolar Disorder in Remission With Signs of Impaired Impulse Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Stare Budgetary Scientific Institution, Mental Health Research Center (Other)
Collaborators: Kazan State Medical University (Other); Federal State Budgetary Institution V.M. Bekhterev National Research Medical Center for Psychiatry and Neurology, Saint-Petersburg, Russia (Unknown)
Responsible Party: Principal Investigator, Margarita Morozova, Head of laboratory of psychopharmacology, PhD,, Federal Stare Budgetary Scientific Institution, Mental Health Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBAD-1
Record Dates: First submitted 2021-09-13; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Bipolar Affective Disorder
Keywords: Bipolar Affective Disorder remission; Impulsivity; Barrat scale; Go-no-go; BART; Ballon Analog Risk Task; Quetiapine
MeSH Terms: conditions — Bipolar Disorder; Impulsive Behavior | interventions — Quetiapine Fumarate

STUDY DESIGN:
Intervention Model Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Quetiapine 25-75 mg (Experimental): There is one arm in this study. Patients will take quetiapine in dose 25-75 1-3 times a day.
  Dose and its frequency can be adjusted by researcher during first 2 weeks (till visit 2), after that patients will take stable dose of quetiapine till week 6 (visit 3).
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — 25-75 mg per day for 6 weeks
  Other Names: Quetiapine - impulsivity

SUMMARY:
In this study, the task was to evaluate the effectiveness of prescribing small doses of quetiapine (25-75 mg) for bipolar patients in remission in order to relieve symptoms of impulsivity.

DETAILED DESCRIPTION:
The purpose of this study is to study the efficacy and safety of the administration of Quetiapine ® in small doses (25-75 mg / day) to patients diagnosed with bipolar disorder who are in an euthymic state with signs of impaired impulse control.

The method of administration, dosage regimen and duration of taking quetiapine in this study: 1-3 tablets from one to 3 times a day, regardless of food intake for 28 days.

Each patient included in the program will be given a package with the drug for 14 days of admission. In the first 14 days of administration, dose adjustment is possible in the range from 25 to 75 mg, depending on individual tolerability. The decision on correction is made by the doctor based on a phone call to the patient after the first week of taking the drug at a dose of 25 mg. Correction is also possible at a later or earlier date during the first two weeks of therapy. At visit 2, the patient will have to provide the doctor with a package of the drug as part of the compliance assessment. At visit 2, the doctor should give the patient packages with the drug for 28 days of admission and ask them to bring packages to assess compliance and account for the drug for visit 3.

Screening (Visit 1 / Day 0) The inclusion of the subject in the program will be carried out on the basis of an assessment of demographic, clinical characteristics, anamnesis data. Prior to the start of the examination, the subject must be provided with oral information about the nature of the study, an informed consent form for signing.

The following procedures will be performed during the screening:

* Collection of demographic data;
* Medical history (previous and concomitant diseases, surgical interventions, allergic history, gynecological history);
* Confirmation of the diagnosis
* Evaluation of inclusion/non-inclusion criteria;

  -- Registration of the drug (or other) therapy that the study participant receives;
* The presence of bad habits;
* Rating on the YMRS scale;
* Assessment on the MADRS scale;
* Assessment on the Barratt impulsivity scale;
* Score on the Go-no-go task
* Score on the Ballon Analog Risk Task (BART)
* Delivery of the drug
* Functional magnetic resonance imaging (fMRI) (optional)

Visit 2 / Day 14±3

The following procedures will be carried out on Visit 2:

* Registration of the drug (or other) therapy that the study participant receives;
* Assessment of the subject's compliance;
* Correction of the dose of the drug*;
* Registration of adverse reactions / adverse events;
* Assessment on the Barratt impulsivity scale;
* Score on the Go-no-go task
* Score on the Ballon Analog Risk Task (BART)
* Delivery of the drug
* fMRI (optional)

Visit 3 / Day 42±3 Registration of the drug (or other) therapy that the study participant receives;

* Assessment of the subject's compliance;
* Registration of adverse reactions / adverse events;
* Assessment on the Barratt impulsivity scale;
* Score on the Go-no-go task
* Score on the Ballon Analog Risk Task (BART)
* fMRI (optional)

Concomitant therapy Within the framework of this study, patients can receive any pharmacotherapy therapy, with the exception of quetiapine in higher doses than prescribed by the protocol. At each visit, the doctor should interview the patient about any medications used by the patient during participation in the study. Information about the patient's intake of concomitant medications is entered by the doctor in the IRC.

Functional magnetic resonance imaging (fMRI) As part of this study, an additional fMRI procedure will be performed for a part of patients (10 people) to assess the functional activity of the brain when performing the Go-no-GO test.

Total duration of the study The expected duration of the subjects' participation in the study corresponds to the expected duration of taking the drug and for each participant will be 42 ± 3 days. The inclusion of patients in the study will continue until their total number reaches 30 people.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of written informed consent to participate in the Program.
2. The established diagnosis of bipolar disorder in incomplete remission and the presence of violations in the field of impulse control (score on the Barratt scale above 70 points)
3. Age from 18 to 65 years inclusive;
4. The patient's desire and ability to participate in the study and follow the doctor's instructions.

Exclusion Criteria:

1. The presence of quetiapine intolerance in the anamnesis.
2. The presence of an actual active phase of bipolar disorder: depression (MADRS score above 22 points) or mania (YMRS score above 20 points).
3. Hypersensitivity to the components of quetiapine in the anamnesis;
4. Current clinically significant and unstable somatic diseases.
5. Participation in other observational programs or clinical trials during the conduct of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Statistically significant changes in Barratt Impulsiveness Scale | 6 weeks of treatment
  Statistically significant changes in Barratt Impulsiveness Scale from visit 1 to visit 3. Minimum score for this scale is 55, maximum score is 120, higher scores mean worse outcome.
Statistically significant changes in total earnings score of Ballon Analog Risk Task (BART) | 6 weeks of treatment
  In Ballon Analog Risk Task (BART) participants should earn as many points as they can during task. Total score is major parameter, measured in points, more points means better outcome.
Statistically significant changes in dprime parameter in Go-no-Go task | 6 weeks of treatment
  In Go-no-Go task participants should push the button on keyboard whan they see certain pictures and dont push when there see any other pictures. Dprime is major parameter which summarizes number of right and wrong answers, measured in points, more points means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Margarita A Morozova, PhD, Principal Investigator — Federal Stare Budgetary Scientific Institution, Mental Health Research Center
Locations (1):
- Mental health research center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No